CLINICAL TRIAL: NCT00919919
Title: Efficacy & Tolerability of Progesterone Vaginal Tablets (Endometrin®) in Menopausal Women Treated by Estrogen Replacement Therapy - Phase II Comparative Study
Brief Title: Efficacy and Tolerability Study of Progesterone Vaginal Tablets (Endometrin®) in Menopausal Women Treated by Estrogen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Prof. Boris Kaplan, Gynecology Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fr003; 5340/09
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Endometrial Hyperplasia; Endometrial Cancer
Keywords: menopause; Endometrial Thickness; progesterone
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Progesterone; estradiol, norethindrone drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone vaginal tablet (Experimental): Group A - Daily use of Endometrin 100 mg progesterone vaginal tablet, and Estrofem orally.
  Interventions: Drug: progesterone
- Activella (Other): Daily use of 1 mg estradiol and 0.5 mg norethindrone acetate administrated orally
  Interventions: Drug: activella

INTERVENTIONS:
Drug: progesterone — Daily use of 100 mg progesterone vaginal tablet, and Estrofem; estradiol 1 mg administrated orally. for 6 month
  Other Names: Endometrin
  Arms: Progesterone vaginal tablet
Drug: activella — Daily use of 1 mg estradiol and 0.5 mg norethindrone acetate administrated orally
  Arms: Activella

SUMMARY:
The objective of the study is to confirm that the efficacy of vaginal progesterone is at least as good as oral progesterone in order to protect the endometrium of uncontrolled proliferation and prevent endometrial cancer.

DETAILED DESCRIPTION:
Estrogen Replacement Therapy must be opposed by progesterone in order to protect the endometrium of uncontrolled proliferation and prevent endometrial cancer, in women with an intact uterus.

ELIGIBILITY:
Inclusion Criteria:

* Women who are candidates for Hormone Replacement Therapy due to menopausal symptoms.
* Women with an intact uterus.
* No menses within the 12 months preceding screening visit and /or FSH >30 IU/L.
* Endometrial thickness ≤ 5 mm.

Exclusion Criteria:

* Submucosal fibroid/s that applying pressure and affecting endometrial thickness
* Other medication that could affect estrogenic state.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-09 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Comparing the proportion of women with endometrial thickness not exceeding 8mm and change not exceeding 3mm between the two groups. | 1 year

SECONDARY OUTCOMES:
Comparison of the proportion of bleeding pattern between the two groups. | 1 year
To demonstrate that vaginal progesterone tablets decrease systemic progesterone adverse reactions using a questionnaire. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Boris Kaplan, prof, Principal Investigator — Rabin Medical Center Beilinson Hospital
Locations (1):
- Rabin Medical Center Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Background] 1. Jennifer Blake. Menopause: evidence-based practice. Best Practice & Research Clinical Obstetrics and Gynaecology. 2006;20:799-839 2. Deborah Graby: Management of Menopausal Symptoms. The NEW ENGLAND JOURNAL of MEDICINE. 2006; 355:2338-47 3. Elena M. Treatment Strategies for Reducing the Burden of Menopause-Associated Vasomotor Symptoms. Journal of Managed Care Pharmacy. 2008;14(3):s14-s19 4. T.Levy. Z.Ben-Refael et al. Pharmacokinetics of natural progesterone administered in the form of a vaginal tablet. Human Reproduction. 1999;14(3):606-10 6. Devroey P, Palermo G, Bourgain C, et al. Progesterone administration in patients with absent ovaries. Int J Fertile. 1989;34:188- 93 7. Maxson WS, Hargrove JT. Bioavailability of oral micronized progesterone. Fertile Steril. 1985;44:622-26 8. C.Ficicioglu, B. Gurbuz, H. Canova. High local endometrial effect of vaginal progesterone gel. Gynecol Endocrinol. 2004;18:240-43 9. Steege JF, Rupp SL, Stout AL, et al. Bioavailability of nasally administered progesterone. Fertile Steril. 1986;46:722-29 10. Chakmakjian ZH, Zachariah NY. Bioavailability of progesterone with different modes of administration. J Reprod Med. 1987;32:443-48